CLINICAL TRIAL: NCT02521636
Title: Clinical Trial Assessing the Value of an Antibiotic Protocol Guided by Serum Procalcitonin in Acute Exacerbations of Chronic Obstructive Pulmonary Disease in Intensive Care
Acronym: BPCTréa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-038
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anibiotic therapy guided with actual french recommandations (Placebo Comparator): Guided by the antibiotic 2006 recommendations of the French consensus conference on anti-infective therapy of respiratory tract infections in low immuno-competent adult.
  Interventions: Other: Antibiotic therapy randomization
- Anibiotic therapy guided with serum PCT value (Experimental): Guided antibiotic therapy serum PCT at admission, revalued at day 1, day 3 and day 6 as long as PCT is not less than 0.1 ng / mL:
  * PCT <0.1 ng / mL: no antibiotics
  * 0.1 <PCT <0.25 ng / mL: antibiotic advised
  * PCT> 0.25 ng / mL: highly recommended antibiotics
  Interventions: Other: Antibiotic therapy randomization; Other: Serum PCT dosage

INTERVENTIONS:
Other: Antibiotic therapy randomization
Other: Serum PCT dosage
  Arms: Anibiotic therapy guided with serum PCT value

SUMMARY:
Investigators propose to conduct a prospective, randomized, controlled, multicenter assessing the interests of an antibiotic protocol guided by serum procalcitonin (PCT) on morbidity and mortality in patients with chronic obstructive pulmonary disease (COPD) hospitalized in intensive care unit (ICU) for acute exacerbation with or without associated pneumonia. The main objective is to show in patients hospitalized in intensive care for acute exacerbation of COPD with or without pneumonia, safety, defined as a lack of difference in mortality at 3 months, an antibiotic strategy guided by the PCT in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years
* Documented or suspected clinically COPD according to the criteria of GOLD
* In acute exacerbation
* Suspect of lower respiratory tract infection
* With or without pulmonary criteria defined as the presence of a radiological infiltrates consistent with an infectious site and associated with one or more of the following items: dyspnea, cough, sputum, fever above 38 ° C, fireplace clinical auscultation, higher leukocytosis at 10,000 / mm³ or leukopenia below 4000 / mm³
* Admitted to the hospital for less than 48 hours
* ICU Admission
* Informed Consent signed by the patient or his representative

Exclusion Criteria:

* Other than acute exacerbation etiology with or without pulmonary disease as suspected cause of ICU admission
* Patient immunocompromised neutropenia neutrophil count below 500 / mm³ secondary to chemotherapy, corticosteroids greater than 0.5 mg / kg / day for more than 10 days, HIV seropositivity
* Severe Acute Asthma
* Moribund patient or a disease with an estimated survival time of less than three months
* Therapeutic limitation Existence
* minor patient or under guardianship or custody
* Pregnant woman
* Refusal to participate in the study
* The inclusion of the subject in another biomedical research protocol in progress or for less than 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
mortality | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Intensive Care Unit, CHU Caen, Caen, France